CLINICAL TRIAL: NCT02168751
Title: STUDY OF PULMONARY AND SYSTEMIC INFLAMMATORY RESPONSE SECONDARY TO LUNG RESECTION SURGERY USING INTRAVENOUS ANESTHESIA VERSUS INHALATION ANESTHESIA WITH HALOGENATED AGENTS
Brief Title: Inflammatory Response Secondary Using Intravenous Anesthesia Versus Inhalation Anesthesia With Halogenated Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIBHGM-ECNC003-2011; 2011-002294-29 (EudraCT Number)
Record Dates: First submitted 2012-07-19; First posted 2014-06-20 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Resection
Keywords: one lung ventilation; inflammatory response; thoracic surgery
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): propofol doses to maintain hypnoses between 40-60 bis(Bispectral Index Scale)during the lung resection surgery
  Interventions: Drug: propofol
- sevoflurane (Experimental): Sevoflurane doses to maintain hypnoses between 40-60 bis(Bispectral Index Scale)during the lung resection surgery
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: propofol
  Arms: propofol
Drug: Sevoflurane
  Arms: sevoflurane

SUMMARY:
Lung ventilation required for lung resection surgery induces a proinflammatory response including cytokine production and recruitment of leukocytes and macrophages in the lung associated with postoperative complications, mainly acute lung injury (ALI). The lung-protective ventilation has been shown reduce this inflammatory response and play a protective role against ALI, even though it is unclear the role of intravenous and inhalational anesthetic agents in immunomodulation of the inflammatory response during lung ventilation and its possible protective role against ALI. This study aims to determine the effect of anesthetic agents on markers of lung inflammation, the mechanisms of oxidative stress and ischemia-reperfusion, and assess the relationship between these mediators and postoperative morbidity defined as percentage of postoperative lung complications (ALI / ARDS, pneumonia and atelectasis), length of stay in ICU, hospital stay and mortality at 30 days. The investigators hypothesis, based on results of our group in animal research, is that inhalants cause a lower proinflammatory response to intravenous agents for lung resection surgery.

A clinical trial is design with two groups (propofol, sevoflurane) managed all with lung protective ventilation, in which the markers will be measured before and after one-lung ventilation in both lungs and in plasma before, during and after one-lung ventilation. postoperative lung complications, ICU and hospital stay and 30 days mortality.

ELIGIBILITY:
Inclusion Criteria:

* candidates to Lung resection surgery at Hospital General Universitario Gregorio Marañón (males and females)
* willing to participate and sign informed consent
* age > 18 años and legal capable
* no urgent surgery.
* FEV1 >50% or CVF > 50%
* no previous steroids or immunosuppressors chronic treatment (three months before the surgery)

Exclusion Criteria:

* pregnancy and breast feeding
* propofol or sevoflurane hypersensibility.
* have received blood derivate product within 10 days before surgery.
* when protective pulmonary ventilation is not possible during one Lung ventilation.
* Heart failure > II NYHA within one week before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in inflammation markers in plasma and bronchoalveolar lavage | baseline and 5 minutes
  Fiberoptic bronchoalveolar lavage (BAL) performed in both lungs at two moments: Baseline ( 5 minutes before the begining of OLV) and at the end of the OLV ( 5 minutes after the two lung vetilation was restored).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco de la Gala, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Anesthesiology Department Hospital GU Gregorio Mrañón, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Alonso A, de la Gala F, Vara E, Hortal J, Pineiro P, Reyes A, Simon C, Garutti I. Lung and blood perioperative metalloproteinases in patients undergoing oncologic lung surgery: Prognostic implications. Thorac Cancer. 2024 Feb;15(4):307-315. doi: 10.1111/1759-7714.15190. Epub 2023 Dec 28. PMID 38155459
- [Derived] Garutti I, De la Gala F, Pineiro P, Rancan L, Vara E, Reyes A, Puente-Maestu L, Bellon JM, Simon C. Usefulness of combining clinical and biochemical parameters for prediction of postoperative pulmonary complications after lung resection surgery. J Clin Monit Comput. 2019 Dec;33(6):1043-1054. doi: 10.1007/s10877-019-00257-4. Epub 2019 Jan 17. PMID 30656507
- [Derived] de la Gala F, Pineiro P, Reyes A, Vara E, Olmedilla L, Cruz P, Garutti I. Postoperative pulmonary complications, pulmonary and systemic inflammatory responses after lung resection surgery with prolonged one-lung ventilation. Randomized controlled trial comparing intravenous and inhalational anaesthesia. Br J Anaesth. 2017 Oct 1;119(4):655-663. doi: 10.1093/bja/aex230. PMID 29121283